CLINICAL TRIAL: NCT02611089
Title: Muscle Connective Tissue in Limb Development and Disease
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14SG01; 15/LO/2085 (Other: London Hampstead REC)
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Radial Dysplasia
Keywords: Muscle connective tissue; Small leucine-rich proteoglycans; Limb development

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue biopsies measuring no more than 5 x 10 mm, consisting of muscle, muscle connective tissue, tendon, fat and skin, or a combination of the above, and / or; Tissue normally discarded during the patient's routine reconstructive hand surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Radial dysplasia patients: Recruited participants will have 2-3 small tissue biopsy samples taken during 1-2 of their planned reconstructive surgical procedures for radial dysplasia, whilst under general anaesthesia in the operating theatre. Samples will be taken by scalpel or scissors, by the operating surgeon, from within the surgical site in the forearm and hand. The skin incision and deep dissection will have to be made as part of the normal course of reconstructive surgery, regardless of participation in this study.
  Interventions: Procedure: Tissue biopsy
- Control patients: Recruited participants will have 2-3 small tissue biopsy samples taken during their planned reconstructive surgery for hand trauma, whilst under general anaesthesia in the operating theatre. Samples will be taken by scalpel or scissors, by the operating surgeon, from within the surgical site in the forearm and hand. The skin incision and deep dissection will have to be made as part of the normal course of reconstructive surgery, regardless of participation in this study.
  Interventions: Procedure: Tissue biopsy

INTERVENTIONS:
Procedure: Tissue biopsy — Sampling of tissue as described.

SUMMARY:
The objective of this work is to understand how the disruption of the muscle connective tissue contributes to the limb soft-tissue defects in radial dysplasia. In parallel, the researchers will investigate the role of muscle connective tissue in normal limb development.

DETAILED DESCRIPTION:
The objective of this work is to understand the origins of the soft tissue defects in a disabling, disfiguring limb anomaly called radial dysplasia, and what mechanisms of normal limb development have been disrupted in these patients to produce their phenotype. The investigators aim to use this knowledge to improve their treatment. Currently, despite sophisticated surgical treatment, the limb malformation the child is born with typically recurs as they grow: it is thus an 'unsolved problem'.

The investigators have previously shown, in an experimental mouse model of radial dysplasia, the underlying soft tissue problem is a change in the muscle connective tissue and its derivatives, causing abnormal soft-tissue patterning. The investigators wish to expand this work into the investigators' patient population by comparing samples of post-natal muscle connective tissue derivatives from radial dysplasia patients with control samples.

The investigators will ask patients undergoing corrective hand surgery to let the investigators take small tissue samples during their planned operations. The investigators will also ask patients having other forms of hand surgery, such as surgery for hand injuries, to let the investigators take similar samples for comparison. In either case, their scar and peri-operative treatment will be unchanged. The investigators will examine the tissue samples in the investigators' laboratory to look for changes in tissue architecture, cellular composition, cell signalling, and how they behave when grown in culture. The investigators will also make attempts to derive cell lines from biopsy samples to use in further studies, exploring cellular phenotype and functional capacity.

Simultaneously, the investigators will look at the long-term surgical outcomes and the range of genetic changes in the investigators' patient population. Eligible patients will be referred for consideration in the (separate) 100,000 genome project; this should further expand the investigators' knowledge of the genetic changes underlying limb anomalies. The ability to combine data on genotype, long-term phenotype and soft tissue changes will give a comprehensive overview of the condition. The investigators expect this to lead to a better understanding of patient subgroups, and to provide a rational basis for improved treatment approaches.

ELIGIBILITY:
Cases

Inclusion Criteria:

* Patients with a clinical diagnosis of radial dysplasia, requiring reconstructive surgery
* Either sex
* Informed (parental) consent to participate

Exclusion Criteria:

* Patients with a clinical diagnosis of radial dysplasia, but not requiring reconstructive surgery
* Patients with a diagnosis other than radial dysplasia
* Patients with extensive previous scarring to their forearm and hand.
* Patients with a significant pathological skin or soft tissue lesion at the donor site.

Controls

Inclusion Criteria:

* Patients with an injury requiring reconstructive surgery
* Either sex
* Informed (parental) consent to participate

Exclusion Criteria:

* Patients with extensive previous scarring to their forearm and hand.
* Patients with a significant pathological skin or soft tissue lesion at the donor site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases - Any patient attending Great Ormond Street Hospital or Guy's and St Thomas' Hospital for reconstructive hand surgery.
  Controls - Any patient attending Great Ormond Street Hospital, Guy's and St Thomas' Hospital Oxford University Hospitals, Chelsea and Westminster or the Royal Free Hospital for reconstructive hand surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-02-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2036-08 (Estimated)

PRIMARY OUTCOMES:
Characterisation of muscle connective tissue derivatives - structure | 3 years
  The characterization of any structural difference in tissue organisation within muscle connective tissue derivatives, comparing normal control patients to patients with radial dysplasia.
Characterisation of muscle connective tissue derivatives - function | 3 years
  The characterization of any functional difference in gene expression within muscle connective tissue derivatives, comparing normal control patients to patients with radial dysplasia.

SECONDARY OUTCOMES:
Identification of biomarker(s). | 3 years
  The identification of a novel biomarker (or biomarkers) for human muscle connective tissue derivatives, which may potentially serve as a diagnostic or prognostic tool
Identification of muscle connective tissue progenitor-cell pool. | 3 years
  The potential identification of a stem-cell-like or progenitor-cell pool for muscle connective tissue derivatives in mature soft tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Logan, PhD, Study Chair — King's College London; Branavan Sivakumar, FRCS(Plast), Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; Gill Smith, FRCS(Plast), Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; George Murphy, PhD FRCS, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; Lucy Cogswell, FRCS(Plas), Principal Investigator — Oxford University Hospitals
Locations (5):
- United Kingdom (5):
  - Oxford University Hospitals, Oxford, Oxfordshire
  - Royal Free Hospital, London
  - Guy's and St Thomas' Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website - for version control & distribution of patient information leaflets / consent forms. — http://congenitalhand.net/

DOCUMENTS (1):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT02611089/Prot_000.pdf